CLINICAL TRIAL: NCT01630473
Title: Clinical Comparison Between the Corticotomy-assisted Orthodontics and Conventional Orthodontics
Brief Title: Effect of Corticotomy on the Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Javier Enrique Botero, Full Time Professor of Periodontics, Universidad de Antioquia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORT2011
Record Dates: First submitted 2012-06-24; First posted 2012-06-28 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Tooth Crowding
Keywords: Tooth crowding; Teeth malpositions; corticotomy; orthodontics; tooth movement; periodontal parameters
MeSH Terms: conditions — Malocclusion | interventions — Osteotomy; Orthodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corticotomy-assisted orthodontics (Experimental): This group of patients will receive corticotomy surgical procedure at day 0. Orthodontic activation will start immediately after surgery.
  Interventions: Procedure: Corticotomy
- Conventional orthodontics (Active Comparator): This group of patients will receive conventional orthodontics starting at day 0.
  Interventions: Procedure: Conventional orthodontics

INTERVENTIONS:
Procedure: Corticotomy — After a periodontal full flap is dissected, by using small round burs, vertical lines (2 mm depth corticotomy) parallel to each root of the teeth in the anterior segment (canines and incisors) are created 5 mm beyond the apex in the maxillary bones and interconnecting the lines at the apex by horizontal corticotomies. Marginal bone crest is not touched by the surgical procedure.
  Other Names: Osteotomy
  Arms: Corticotomy-assisted orthodontics
Procedure: Conventional orthodontics — Conventional orthodontic treatment
  Other Names: Orthodontic treatment
  Arms: Conventional orthodontics

SUMMARY:
Orthodontic therapy allows for the treatment of dental malpositions in order to produce an adequate relationship between teeth during occlusion. Conventional orthodontic therapy applies slight forces and moves teeth slowly. It is generally performed during a 2 year minimum of time. Recent studies seem to suggest that orthodontic therapy time can be shortened by surgical assistance (corticotomy). This investigation is aimed to determine the velocity of tooth movement and changes in periodontal clinical parameters between corticotomy-assisted orthodontic therapy and conventional orthodontic therapy.

DETAILED DESCRIPTION:
The use of surgical techniques to accelerate orthodontic tooth movement has been developed. By means of surgical burs, vertical grooves in the cortical plate (corticotomy) are produced mesial and distal to the roots of teeth that are being moved 3 mm below the marginal crest and extending beyond the apex. Animal studies showed that the rapid orthodontic tooth movement was due to increased cellular activity in the surrounding periodontal tissues, a regional acceleratory phenomenon (RAP). A high osteoclastic activity is observed in the compression side although is also observed in the tension side to a less degree. Histological analysis indicates that at day 21 the remodeling tissues are replaced by a fibrous tissue and later (60 days) by bone. Furthermore, the tissues immediately adjacent to the corticotomy are characterized by an increased width of the periodontal ligament, less calcified spongiosa bone surface and higher counts of osteoclasts. But not only the catabolic activity is increased (osteoclasts) but also the anabolic activity (osteoblasts) is increased 3-fold as well. This balances the rate of bone resorption and bone apposition. An interesting finding was the reduced rate of hyalinization at the compression site, which may be due to increased width of the periodontal ligament and thus facilitating tooth movement.

As opposed to conventional osteotomy used in alveolar distraction, the preservation of the medullar vasculature during a corticotomy procedure provides and adequate blood supply and nutrition. This accelerates the rate of tissue healing and remodeling and hence orthodontic movement can start immediately after surgery. It has been calculated that the rate of tooth movement is doubled (2.5mm to 3mm at day 25) in comparison to standard orthodontics without any detrimental effects on periodontal tissues. This surgically assisted approach for improved tooth movement is beneficial for molar intrusion, space closure, de-crowding and open bite management.

This investigation is aimed to determine the velocity of tooth movement and changes in periodontal clinical parameters between corticotomy-assisted orthodontic therapy and conventional orthodontic therapy. Periodontally and systemically healthy subjects in need of orthodontic therapy for the treatment of teeth crowding in the anterior segment. The rate of tooth movement will be assessed by radiographs and cast models and periodontal clinical parameters will be recorded at each visit during the 4 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation
* Legally adult age (>18 years old)
* Full permanent dentition (28 teeth excluding third molars)
* Severe anterior teeth crowding
* Thick periodontal biotype

Exclusion Criteria:

* Systemic diseases (i.e. diabetes, HIV)
* cigarette smoking
* Under medications: bisphosphonates, anti-epileptic drugs, contraceptives, corticosteroids, estrogen, antihistamine drugs, calcitonin, vitamin D
* Previous orthodontic treatment
* Periodontal disease
* Severe gingival recessions
* Pregnancy
* Previous root resorption

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes in tooth position | 0 days, 7 days, 15 days, 1st month, 2nd month, 3rd month and 4th month after surgery and conventional orthodontic

SECONDARY OUTCOMES:
Periodontal Clinical Parameters | 0 days, 7 days, 15 days, 1st month, 2nd month, 3rd month and 4th month after surgery and conventional orthodontic

CONTACTS AND LOCATIONS:
Overall Officials: Juan D Arango, DDS, Principal Investigator — Faculty of Dentistry, Universidad de Antioquia; Javier E Botero, PhD, Study Director — Faculty of Dentistry, Universidad de Antioquia
Locations (1):
- Faculty of Dentistry, Universidad de Antioquia, Medellín, Antioquia, Colombia

REFERENCES:
- [Background] Nowzari H, Yorita FK, Chang HC. Periodontally accelerated osteogenic orthodontics combined with autogenous bone grafting. Compend Contin Educ Dent. 2008 May;29(4):200-6; quiz 207, 218. PMID 18533317
- [Background] Wilcko WM, Wilcko T, Bouquot JE, Ferguson DJ. Rapid orthodontics with alveolar reshaping: two case reports of decrowding. Int J Periodontics Restorative Dent. 2001 Feb;21(1):9-19. PMID 11829041
- [Background] Ozturk M, Doruk C, Ozec I, Polat S, Babacan H, Bicakci AA. Pulpal blood flow: effects of corticotomy and midline osteotomy in surgically assisted rapid palatal expansion. J Craniomaxillofac Surg. 2003 Apr;31(2):97-100. doi: 10.1016/s1010-5182(02)00188-9. PMID 12628599
- [Background] Koudstaal MJ, Wolvius EB, Schulten AJ, Hop WC, van der Wal KG. Stability, tipping and relapse of bone-borne versus tooth-borne surgically assisted rapid maxillary expansion; a prospective randomized patient trial. Int J Oral Maxillofac Surg. 2009 Apr;38(4):308-15. doi: 10.1016/j.ijom.2009.02.012. Epub 2009 Mar 10. PMID 19278832
- [Background] Akay MC, Aras A, Gunbay T, Akyalcin S, Koyuncue BO. Enhanced effect of combined treatment with corticotomy and skeletal anchorage in open bite correction. J Oral Maxillofac Surg. 2009 Mar;67(3):563-9. doi: 10.1016/j.joms.2008.06.091. PMID 19231781